CLINICAL TRIAL: NCT05279690
Title: Colchicine to Suppress Pro-tumorigenic Inflammation in Patients with Urothelial Cancer and Other Solid Tumors
Brief Title: Pilot Trial of Colchicine in Urothelial Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Deborah Doroshow, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01175
Record Dates: First submitted 2022-03-05; First posted 2022-03-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Cancer; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 low-dose colchicine (Experimental): Participants with advanced/recurrent solid tumors who will receive low-dose colchicine (0.6 mg oral BID)
  Interventions: Drug: Colchicine
- Cohort 1 high-dose colchicine (Experimental): Participants with metastatic solid tumors who will receive high-dose colchicine (0.6 mg oral TID)
  Interventions: Drug: Colchicine
- Cohort 2 Participants with post-radical surgery (Experimental): Participants with post-radical surgery for high-risk clinically localized urothelial cancer will receive colchicine 0.6 mg oral BID.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Patients will receive 14 days of colchicine in the absence of prohibitive toxicity of disease progression

SUMMARY:
This open-label, non-randomized study aims to determine the anti-inflammatory effect of colchicine on the reduction of peripheral blood CRP in patients with solid tumors or localized urothelial cancer. There are two cohorts, which will enroll separately and parallelly. Cohort 1 will include two successive groups with advanced/recurrent solid tumors (15 patients will receive low-dose colchicine and 15 for high-dose colchicine) who will receive 14 days of colchicine. In Cohort 2, 15 patients with post-radical surgery for high-risk clinically localized urothelial cancer will be enrolled. They will receive one 28-day cycle of colchicine. The primary outcome, post-treatment decline in CRP level, a continuous measure, will be defined as the maximum percentage decline from baseline in post-treatment CRP value within two weeks of colchicine (Cohort 1) or one cycle of colchicine (cohort 2), where the baseline value is measured before any treatment is initiated.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration. ECOG 2 is allowed for patients on Cohort 1.
* Cohort 1:

  * Histological or cytologically confirmed solid tumor.
  * Metastatic or recurrent disease
  * Elevated peripheral blood CRP level (> 5 mg/L) documented on routine bloodwork within 14 days or registration.
* Cohort 2:

  * History of urothelial cancer post radical cystectomy, nephroureterectomy, or ureterectomy
  * Eligible and planned for standard of care adjuvant nivolumab in the opinion of the treating investigator
  * Elevated peripheral blood CRP level (> 5 mg/L) documented on routine bloodwork at a minimum of 30 days and a maximum of 120 days after surgical resection and within 14 days prior to registration.
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks preferred) or at least 15 unstained slides. If archival tissue is not available, enrollment will be considered on a case by case basis after discussion with the Principal Investigator.
* Demonstrate adequate organ function as defined below. All screening labs to be obtained within 14 days prior to registration.

  * White blood cell (WBC) ≥ 2.5 K/mm3
  * Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
  * Hemoglobin (Hgb) ≥ 8 g/dL
  * Calculated GFR ≥ 50 cc/min or creatinine ≤ 1.5 mg/dl (The CKD-EPI equation will be used to calculate GFR)
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN or < 5xULN for patients in Cohort 1 with liver metastases
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN or < 5xULN for patients in Cohort 1 with liver metastases
* Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. See section 5.5 for definition of childbearing potential.
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use an effective method(s) of contraception from the time of informed consent, during the study until after the last dose of study drug(s). Males must be willing to abstain from heterosexual activity or to use an effective method(s) of contraception from initiation of treatment until after the last dose of study drug(s).
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* Patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

* Already taking long term colchicine for any other reason.
* Active infection requiring systemic therapy.
* Pregnant or breastfeeding.
* Prior cancer treatment must be completed at least 30 days prior to registration, or within 5 half-lives, and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to Grade ≤ 1 or baseline.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion, are not eligible for this trial.
* Active central nervous system (CNS) metastases.
* Treatment with any investigational drug within 30 days prior to registration.
* Need for concomitant treatment with moderate or strong CYP3A4 inhibitors or P-gp inhibitors.
* Rheumatoid arthritis, vasculitis, systemic lupus erythematosus, or other autoimmune condition requiring active systemic treatment.
* Myocardial infarction within the prior last 6 months and/or ≥ Class III New York Heart Association heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Percent Change in Peripheral blood CRP level | Baseline and Within 28 days
  The primary outcome, post-treatment decline in peripheral blood CRP level, a continuous measure, will be defined as the maximum percent decline of post-treatment CRP from baseline obtained during the treatment period, where the baseline value is measured before any treatment initiated For a patient with an advanced/recurrent solid tumor who receive 2-weeks of treatment, it will be the maximum percentage decline during the 28 days of treatment. For a patient who receive colchicine less than 28 days, it will be the maximum percentage decline from baseline to the last day of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Doroshow, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to the small cohort size.